CLINICAL TRIAL: NCT00850278
Title: Assessment of [18F]FLT-PET Imaging for Diagnosis and Prognosis of Brain Tumors
Acronym: FLT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Collaborators: National Cancer Institute, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2007-006265-32
Record Dates: First submitted 2009-02-23; First posted 2009-02-24 (Estimated); Last update posted 2012-09-03 (Estimated); Status verified 2012-08

CONDITIONS: Cancer; Brain Tumors
Keywords: Brain tumor; [18F]FLT; [11C]MET; TEP-imaging; tumor cell proliferation
MeSH Terms: conditions — Neoplasms; Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- FLT-PET imaging (Experimental): Prior to surgical resection, patient will undergo [11C]MET PET imaging, [18F]FLT PET imaging, MRI, and spectroscopy imaging.
  Interventions: Other: FLT-PET imaging

INTERVENTIONS:
Other: FLT-PET imaging — Prior to surgical resection, patient will undergo [11C]MET PET imaging, [18F]FLT PET imaging, MRI, and spectroscopy imaging.

SUMMARY:
The primary objective of this study is to assess the efficacy of the radiopharmaceutical 3'-deoxy-3'-[F-18]fluorothymidine, [F-18]FLT, a tracor of cell proliferation, using Positron Emission Tomography (PET) imaging for the tumor diagnosis and prognosis in a group of 50 patients with different type of brain tumors.[F-18]FLT PET imaging will be compared to the current used imaging techniques of MRI, spectroscopy imaging, PET imaging using [11C]MET tracer, immunohistochemical analysis and clinical parameters.

ELIGIBILITY:
Inclusion Criteria:

* adults aged between 18 and 70 years
* must have operable grade II, III or IV glioma, recurrent high grade glioma or brain metastases
* KPS >= 70%
* must have the understanding and ability to sign an informed consent document
* must have adequate liver and kidney function
* be male or non-pregnant, non-lactating females
* patients who are fertile must agree to use an effective method of contraception during participation in the study
* the following laboratory results : absolute neutrophil count >= 1500 cells/µl, platelet count >= 100000 cells/µl, SGOT <= 2.5 x ULN, serum creatinine <= 1.5 x ULN.

Exclusion Criteria:

* contraindication to surgery
* concomitant radio-, chemo-, or immunotherapy
* history of significant dementia
* known diagnosis of Human Immunodeficiency Virus (HIV) infection
* patient with hepatitis B or C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-10; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
To evaluated the aggressive potential of brain tumors related to cell proliferation index measured by [18F]FLT | Day 10

SECONDARY OUTCOMES:
To compare the efficiency of [18F]FLT with [11C]MET | Day 15
To define relations between [18F]FLT uptake and clinical, histological and radiological parameters | Day 90
To define relations between [18F]FLT uptake and patient survival | J90

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Sébastien Guillamo, MD, PhD, Principal Investigator — University Hospital, Caen; Jean-Michel Derlon, Pr, Study Director — University Hospital, Caen
Locations (1):
- Caen University Hospital, Caen, France